CLINICAL TRIAL: NCT01856959
Title: Response of Asthmatic Children's Lung Function to Nebulized Magnesium Sulfate After Acetylcholine Provocation Test: a Clinical Trail
Brief Title: Lung Function Changes of Induced Asthma Children Treated With Inhaled MgSO4
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Dai Jihong, professor, Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MS-2013CQ
Record Dates: First submitted 2013-05-14; First posted 2013-05-20 (Estimated); Last update posted 2013-05-20 (Estimated); Status verified 2013-05

CONDITIONS: Asthma
Keywords: magnesium sulfate; nebulized; lung function
MeSH Terms: conditions — Asthma | interventions — Magnesium Sulfate; Albuterol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- nebulized magnesium sulfate (Experimental): nebulized magnesium sulfate 150mg and consisted about 5 min,which used only once
  Interventions: Drug: Magnesium Sulfate
- nebulized magnesium sulfate & albuterol (Experimental): nebulized magnesium sulfate 150mg & albuterol 2.5mg and consisted about 5 min,which used only once
  Interventions: Drug: magnesium sulfate & albuterol
- nebulized albuterol (Active Comparator): nebulized albuterol 2.5mg and consisted about 5 min,which used only once
  Interventions: Drug: Albuterol

INTERVENTIONS:
Drug: Magnesium Sulfate — 2ml of 7.5% solution of isotonic magnesium heptahydrate, 150 mg
  Arms: nebulized magnesium sulfate
Drug: magnesium sulfate & albuterol — 0.5ml of albuterol mixed with 2ml of isotonic magnesium sulfate,150mg+2.5mg
  Arms: nebulized magnesium sulfate & albuterol
Drug: Albuterol — 0.5ml of albuterol mixed with 1.5cc of normal saline, 2.5 mg
  Arms: nebulized albuterol

SUMMARY:
As a non-selective bronchodilator, magnesium sulfate (MgSO4) is effective when administered intravenously in the treatment of the patients with acute severe asthma not responding to conventional therapy (oxygen, nebulized salbutamol, and corticosteroids), which can resulted in earlier improvement in clinical signs and symptoms of asthma and PEF. However, the use of intravenous MgSO4 administered is not common in clinical practice, because it's prone to have adverse effects and side effects such as nausea, vomiting, facial flushing, hypotension, decreased tendon reflexes and so on with this treatment. The aerosolised route offers the advantage of lower dosage, a shorter time of drug being delivered to the airway smooth muscle and lower incidence of side effects when compared to the intravenous route. At present, there are only a few studies about the effects of nebulized MgSO4 in the treatment of acute asthma in children, and the conclusions are controversial.

ELIGIBILITY:
Inclusion Criteria:

* known cases of controlled bronchial asthma
* ≧4 years of age
* the result was positive after acetylcholine provocation test in follow-up visit

Exclusion Criteria:

* had received corticosteroids (inhaled or systemic) or β2-agonists or theophyllines before the clinic day
* had fever (axillary temperature>38.5℃)
* history of chronic disease like bronchopulmonary dysplasia or cystic fibrosis
* history of renal insufficiency and known allergy to acetylcholine, albuterol or magnesium

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 330 (Actual)
Dates: Start 2011-11; Primary Completion 2013-03 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
changes of lung function after interventions | 10 min and 20 min post-dose
  to observe the changes of the lung function indices(FEV1、PEF) at 10 min and 20 min after inhaling magnesium sulfate, albuterol, or combination of magnesium sulfate and albuterol respectively.

SECONDARY OUTCOMES:
effectiveness of nebulized magnesium sulfate alone | 10 min and 20 min post-dose
  to observe the changes of the lung function indices(FEV1、PEF) at 10 min and 20 min after inhaling magnesium sulfate alone,and compared it with the patients who was nebulized inhalation albuterol alone.
the number of patients with adverse events as a measure of safety and tolerability | 20 min
  to observe if any patient appear side effects or adverse effects like nausea, vomiting, hypotension or the change of deep tendon reflexes et al.

CONTACTS AND LOCATIONS:
Overall Officials: Jihong Dai, M.D., Study Director — Chongqing Medical University
Locations (1):
- Center of Respiratory Disorders,Children's Hospital,Chongqing Medical University, Chongqing, Chongqing Municipality, China